CLINICAL TRIAL: NCT02717949
Title: Oral Hepatitis C Treatment for Indolent Lymphoma (OPTImaL) Study
Acronym: Optimal
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: failure to recruit
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 042015-086
Record Dates: First submitted 2015-11-10; First posted 2016-03-24 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Liver Disease
Keywords: hepatitis C; low-grade lymphoma
MeSH Terms: conditions — Liver Diseases; Hepatitis C; Lymphoma, Non-Hodgkin | interventions — ledipasvir, sofosbuvir drug combination; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sofosbuvir/ledipasvir (Experimental): sofosbuvir and ledipasvir fixed dose combination given orally once a day for genotype 1 and 4.
  Interventions: Drug: sofosbuvir/ledipasvir
- sofosbuvir and ribavirin (Experimental): Sofosbuvir 400 mg given orally once a day with weight-base ribavirin of 1200 mg for those >75 kg and 1000 mg for those <75kg given in divided dose twice a day. This intervention is for genotype 2 and 3
  Interventions: Drug: sofosbuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: sofosbuvir/ledipasvir — sofosbuvir ledipasvir fixed dose combination given once a day by mouth
  Other Names: Harvoni
  Arms: sofosbuvir/ledipasvir
Drug: sofosbuvir — sofosbuvir 400 mg given one a daily orally and weight-based ribavirin given twice a day orally
  Other Names: sovaldi
  Arms: sofosbuvir and ribavirin
Drug: Ribavirin — ribavirin 1200 mg given orally in divided dose for those >75kg and 1000 mg in divided dose for those <75 kg.
  Other Names: copegus; rebetol; ribasphere
  Arms: sofosbuvir and ribavirin

SUMMARY:
There still remains the question if hepatitis C eradication with all oral therapy will lead to a regression or cure of the low grade lymphoma. Thus, the hypothesis of this study is that oral HCV therapy will lead to a high rate of hepatitis C eradication which will correlate with a reduction of the size and extent of low-grade lymphoma. The hypothesis of this study is that subjects with hepatitis C,regardless of genotype, who have low grade lymphoma, when treated for hepatitis C without pegylated interferon will have a regression of low grade non-Hodgkin's lymphoma. In this pilot study we will evaluate the effect of Sofosbuvir/ledipasvir or sofosbuvir/ribavirin based antiviral therapy on the course of a subset of HCV-related low grade B cell non-Hodgkin's lymphoma

Primary Objective This study will assess the safety, as measured by adverse events, in subjects receiving hepatitis C treatment.

Secondary Objective The secondary objective of this study is to assess the rate of overall response of B cell non-Hodgkin's lymphoma defined as either as partial response or complete response according to revised international working group criteria for non-Hodgkin lymphoma.

Primary Endpoint Safety and tolerability of sofosbuvir/ledipasvir or sofosbuvir/ribavirin in subjects with B-cell non-Hodgkin's lymphoma will be assessed by number of adverse events and serious adverse events. In addition, the study will assess the number of subjects who had to stop treatment due to adverse events or serious adverse events. The study will also examine the number of subjects in which treatment for lymphoma had to be given due to clinical progression.

Secondary Endpoints The secondary endpoint(s) of this study is to (1) Assess the rate of overall response of B-cell Non-Hodgkin's lymphoma defined as either as partial response or complete response according to revised international working group criteria for non-Hodgkin lymphoma. (2) Determine the rate of sustained viral response in subjects with low-grade lymphoma.

DETAILED DESCRIPTION:
Methods and Study Design

The study will plans to enroll approximately 21 subjects over the next 6-12 months for this study.

Subjects with low grade lymphoma with confirmed diagnosis of hepatitis C with a viral load > 1000 will be included in this study. Subjects may be treatment naïve or experienced to hepatitis C therapy, however subjects must be treatment naïve to non-Hodgkin's lymphoma treatment to be included in this study. All subjects will undergo staging studies at the time of study screening which will include a whole body scans and a bone marrow biopsy. In those with a prior bone marrow biopsy, those who had bone marrow involvement and biopsy was <3 months from screening, then an additional biopsy is not needed. If bone marrow biopsy did not show bone marrow involvement, a repeat bone marrow biopsy is needed at screening. If complete data is not available from a prior biopsy, a repeat bone marrow biopsy will need to be done. In addition, patients will have staging of liver disease by serologic markers of liver inflammation, such as aspartate aminotransferase (AST) to platelet ratio (APRI) and FibroTest® or (Fibro Sure®) or FibroScan®. If these methods are inconclusive, then a liver biopsy may be obtained to determine if the patient has cirrhosis. Patients will be treated regardless of stage of fibrosis. The rationale for examining cirrhosis is that these patients may not respond as well and will require further surveillance for hepatocellular cancer every 6 months. Additionally, hepatitis C viral load and genotype will be determined prior to initiation of hepatitis C treatment.

Setting:

This will be a multi- center study conducted at University of Texas Southwestern Medical Center, Cornell Medical Center, and Memorial Sloan Kettering Cancer Center. Each site would be expected to enroll 7 subjects in 6-12 months.

Treatment

Genotype 1:

Treatment Naïve, with or without cirrhosis: sofosbuvir/ledipasvir one pill once a day for 12 weeks.

Treatment experienced, with cirrhosis: sofosbuvir/ledipasvir one pill once a day with weight-based ribavirin for 12 weeks. Weight-based ribavirin refers to use 1200 mg of ribavirin in divided doses for those ≥75 kg and 1000 mg in divided dose for those <75kg.

Treatment experienced with cirrhosis : sofosbuvir/ledipasvir one pill once a day for 24 weeks. This option is for subjects who are unable to take ribavirin.

Genotype 2:

Treatment naïve or experienced without cirrhosis: sofosbuvir 400mg once daily and ribavirin 1000/1200 mg weight-based dosing in divided dose twice a day for 12 weeks.Treatment naïve or experienced with cirrhosis: sofosbuvir 400 mg and weight-based ribavirin for 16 weeks

Genotype 3:

Treatment naïve, non-cirrhotic: sofosbuvir/ledipasvir fixed dose combination combined with weight-based ribavirin for 12 weeks or treatment naïve with cirrhosis: sofosbuvir 400 mg daily with weight-based ribavirin for 24 weeks.

Treatment experienced with cirrhosis will be excluded as the best treatment for this population would require pegylated interferon.

Genotype 4:

Treatment naïve with or without cirrhosis or treatment experienced without cirrhosis: sofosbuvir/Ledipasvir fixed dose combination for 12 weeks.

Treatment experienced with cirrhosis: sofosbuvir/ledipasvir for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Male or female >18 years of age
3. Serum HCV RNA levels of >1,000 IU per milliliter or higher
4. HCV treatment experienced or naïve.

   * HCV treatment naïve: No prior exposure to any Interferon, ribavirin, or other approved or experimental HCV-specific directly acting antivirals
   * HCV Treatment-Experienced: Virologic failure after treatment with Pegylated interferon + ribavirin, Non-structural 3/4a (NS3/4A) protease inhibitor plus pegylated interferon + ribavirin, or regimen of sofosbuvir±ribavirin± pegylated interferon regimen.
5. Chronic Hepatitis C based on the judgment of the investigator
6. HCV genotype 1, 2, 3, 4
7. If the patient is determined to be cirrhotic (based on criteria outlined earlier), the patient must have an ultrasound done within 6 months prior to enrollment with no evidence of hepatocellular carcinoma.
8. Indolent Non-Hodgkin's lymphoma , which may include the following :

   * Nodal Marginal zone lymphoma
   * Extranodal marginal zone lymphoma (MALT)
   * Splenic marginal zone lymphoma
   * Follicular lymphoma Grade 1-3a with low tumor burden*, FLIPI 2 risk category of either low (i.e. no risk factors) or intermediate (1-2 risk factors), and with no B symptoms. B symptoms are defined as:

     * Fever (i.e., temperature >38°C [>100.4°F]) for 3 consecutive days
     * Weight loss exceeding 10% of body weight in 6 months
     * Drenching night sweats
   * Lymphoplasmacytic lymphoma
9. No prior chemotherapy

   * Low tumor burden is defined as normal lactate dehydrogenase, largest nodal or extranodal mass less than 7 cm, up to three nodal sites containing nodes with a diameter greater than 3 cm, no clinically significant serous effusions detectable by physical examination or positron emission tomography (PET)/CT scan, and spleen enlargement up to 16 cm by CT without any evidence of portal hypertension.
10. Karnofsky performance status > 70%
11. Creatinine clearance ≥60 mL/min, as calculated by Cockcroft-Gault equation
12. If patient will need ribavirin in their regimen then the following inclusion:

    * Hg >12 g/dL for male
    * Hg >11 g/dL for female
13. All women of child-bearing potential who take ribavirin will need to have a negative urine pregnancy test.

Exclusion Criteria:

1. Life expectancy < 6 months
2. Any HCV treatment which uses pegylated interferon
3. HCV genotype 3 Treatment experienced with cirrhosis
4. Co-infection with hepatitis B
5. Prior chemotherapy for lymphoma
6. Lymphomas of other histologies other than the ones listed in section 3.3 above
7. Follicular lymphoma with large cell transformation
8. Decompensated liver disease in which pegylated interferon is contraindicated.
9. Female who is pregnant or breast feeding and HCV treatment requires use of ribavirin.
10. Solid organ transplant
11. Any interferon- containing agent within 8 weeks prior to screening or any prior exposure to HCV-specific antivirals agent(s), other than NS3/ 4A protease inhibitor and sofosbuvir
12. Known hypersensitivity to ledipasvir, sofosbuvir, or formulation excipients.
13. On a prohibited medication which cannot be stopped during the duration of HCV treatment.
14. Female subject who is pregnant or breastfeeding
15. HIV-infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mamta K. Jain, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (3):
- United States (3):
  - Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Forghieri F, Luppi M, Barozzi P, Maffei R, Potenza L, Narni F, Marasca R. Pathogenetic mechanisms of hepatitis C virus-induced B-cell lymphomagenesis. Clin Dev Immunol. 2012;2012:807351. doi: 10.1155/2012/807351. Epub 2012 Jul 11. PMID 22844326
- [Background] Peveling-Oberhag J, Arcaini L, Hansmann ML, Zeuzem S. Hepatitis C-associated B-cell non-Hodgkin lymphomas. Epidemiology, molecular signature and clinical management. J Hepatol. 2013 Jul;59(1):169-77. doi: 10.1016/j.jhep.2013.03.018. Epub 2013 Mar 27. PMID 23542089
- [Background] Arcaini L, Merli M, Volpetti S, Rattotti S, Gotti M, Zaja F. Indolent B-cell lymphomas associated with HCV infection: clinical and virological features and role of antiviral therapy. Clin Dev Immunol. 2012;2012:638185. doi: 10.1155/2012/638185. Epub 2012 Aug 26. PMID 22956970
- [Background] Kasama Y, Mizukami T, Kusunoki H, Peveling-Oberhag J, Nishito Y, Ozawa M, Kohara M, Mizuochi T, Tsukiyama-Kohara K. B-cell-intrinsic hepatitis C virus expression leads to B-cell-lymphomagenesis and induction of NF-kappaB signalling. PLoS One. 2014 Mar 20;9(3):e91373. doi: 10.1371/journal.pone.0091373. eCollection 2014. PMID 24651473
- [Background] Hermine O, Lefrere F, Bronowicki JP, Mariette X, Jondeau K, Eclache-Saudreau V, Delmas B, Valensi F, Cacoub P, Brechot C, Varet B, Troussard X. Regression of splenic lymphoma with villous lymphocytes after treatment of hepatitis C virus infection. N Engl J Med. 2002 Jul 11;347(2):89-94. doi: 10.1056/NEJMoa013376. PMID 12110736
- [Background] Vallisa D, Bernuzzi P, Arcaini L, Sacchi S, Callea V, Marasca R, Lazzaro A, Trabacchi E, Anselmi E, Arcari AL, Moroni C, Berte R, Lazzarino M, Cavanna L. Role of anti-hepatitis C virus (HCV) treatment in HCV-related, low-grade, B-cell, non-Hodgkin's lymphoma: a multicenter Italian experience. J Clin Oncol. 2005 Jan 20;23(3):468-73. doi: 10.1200/JCO.2005.06.008. PMID 15659492
- [Background] Arcaini L, Vallisa D, Rattotti S, Ferretti VV, Ferreri AJM, Bernuzzi P, Merli M, Varettoni M, Chiappella A, Ambrosetti A, Tucci A, Rusconi C, Visco C, Spina M, Cabras G, Luminari S, Tucci M, Musto P, Ladetto M, Merli F, Stelitano C, d'Arco A, Rigacci L, Levis A, Rossi D, Spedini P, Mancuso S, Marino D, Bruno R, Baldini L, Pulsoni A. Antiviral treatment in patients with indolent B-cell lymphomas associated with HCV infection: a study of the Fondazione Italiana Linfomi. Ann Oncol. 2014 Jul;25(7):1404-1410. doi: 10.1093/annonc/mdu166. Epub 2014 May 5. PMID 24799461
- [Background] Afdhal N, Zeuzem S, Kwo P, Chojkier M, Gitlin N, Puoti M, Romero-Gomez M, Zarski JP, Agarwal K, Buggisch P, Foster GR, Brau N, Buti M, Jacobson IM, Subramanian GM, Ding X, Mo H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Mangia A, Marcellin P; ION-1 Investigators. Ledipasvir and sofosbuvir for untreated HCV genotype 1 infection. N Engl J Med. 2014 May 15;370(20):1889-98. doi: 10.1056/NEJMoa1402454. Epub 2014 Apr 11. PMID 24725239
- [Background] Gane EJ, Stedman CA, Hyland RH, Ding X, Svarovskaia E, Symonds WT, Hindes RG, Berrey MM. Nucleotide polymerase inhibitor sofosbuvir plus ribavirin for hepatitis C. N Engl J Med. 2013 Jan 3;368(1):34-44. doi: 10.1056/NEJMoa1208953. PMID 23281974
- [Background] Kowdley KV, Gordon SC, Reddy KR, Rossaro L, Bernstein DE, Lawitz E, Shiffman ML, Schiff E, Ghalib R, Ryan M, Rustgi V, Chojkier M, Herring R, Di Bisceglie AM, Pockros PJ, Subramanian GM, An D, Svarovskaia E, Hyland RH, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Pound D, Fried MW; ION-3 Investigators. Ledipasvir and sofosbuvir for 8 or 12 weeks for chronic HCV without cirrhosis. N Engl J Med. 2014 May 15;370(20):1879-88. doi: 10.1056/NEJMoa1402355. Epub 2014 Apr 10. PMID 24720702
- [Background] Lawitz E, Poordad FF, Pang PS, Hyland RH, Ding X, Mo H, Symonds WT, McHutchison JG, Membreno FE. Sofosbuvir and ledipasvir fixed-dose combination with and without ribavirin in treatment-naive and previously treated patients with genotype 1 hepatitis C virus infection (LONESTAR): an open-label, randomised, phase 2 trial. Lancet. 2014 Feb 8;383(9916):515-23. doi: 10.1016/S0140-6736(13)62121-2. Epub 2013 Nov 5. PMID 24209977
- [Background] Zeuzem S, Dusheiko GM, Salupere R, Mangia A, Flisiak R, Hyland RH, Illeperuma A, Svarovskaia E, Brainard DM, Symonds WT, Subramanian GM, McHutchison JG, Weiland O, Reesink HW, Ferenci P, Hezode C, Esteban R; VALENCE Investigators. Sofosbuvir and ribavirin in HCV genotypes 2 and 3. N Engl J Med. 2014 May 22;370(21):1993-2001. doi: 10.1056/NEJMoa1316145. Epub 2014 May 4. PMID 24795201

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sofosbuvir/Ledipasvir | Sofosbuvir and Ribavirin
Started (data not reported due to confidentiality) | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: no patients were analyzed due to insufficient numbers and risk of identifying patient by reporting data on 1 person
Groups:
- Total: Total of all reporting groups
Arm/Group | Sofosbuvir and Ribavirin | Sofosbuvir/Ledipasvir | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number Subjects Who Experience Adverse Events on HCV Treatment as Assessed by Division of AIDS (DAIDS) Adverse Event (AE) Grading Table Version 2.0.
Description: number of subjects who experience treatment-related adverse event on HCV treatment as assessed by DAIDS AE Grading Table version 2.
Time Frame: from drug dispensation until post-treatment week 36
Population: data not reported due to confidentiality
Arm/Group | Sofosbuvir/Ledipasvir | Sofosbuvir and Ribavirin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Subjects Who Have a Change in Lymph Node Size From Baseline After HCV Treatment
Description: Number of subjects who have a change in the size of lymph node size from baseline
Time Frame: from baseline to post-treament week 36
Population: data not reported due to confidentiality
Arm/Group | Sofosbuvir and Ribavirin | Sofosbuvir/Ledipasvir
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: data not reported due to confidentiality
Arm/Group | Sofosbuvir/Ledipasvir | Sofosbuvir and Ribavirin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT02717949/Prot_SAP_000.pdf